CLINICAL TRIAL: NCT06419634
Title: Phase I Multicenter, Open-Label, First-in-Human Study of BMS-986497 (ORM-6151) as a Monotherapy, in Double Combination With Azacitidine and in Triple Combination With Azacitidine and Venetoclax in Subjects With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Study of BMS-986497 (ORM-6151) as a Monotherapy, in Double and Triple Combination With Azacitidine and Venetoclax in Participants With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA235-0001; 2024-519537-29 (Other: EU CTR)
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: BMS-986497; First-in-Human; ORM-6151; Acute myeloid leukemia (AML); Myelodysplastic syndrome (MDS); Cluster of differentiation 33 (CD33); G1 to S phase transition 1 (GSPT1); Open label study
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation BMS-986497 (Monotherapy) (Experimental)
  Interventions: Drug: BMS-986497
- Part 2, Cohort A: Dose Expansion BMS-986497 (Combination Therapy) (Experimental)
  Interventions: Drug: BMS-986497; Drug: Azacitidine
- Part 2, Cohort B: Dose Expansion BMS-986497 (Triple Combination Therapy) (Experimental)
  Interventions: Drug: BMS-986497; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: BMS-986497 — Specified dose on specified days
  Other Names: ORM-6151
Drug: Azacitidine — Specified dose on specified days
  Arms: Part 2, Cohort A: Dose Expansion BMS-986497 (Combination Therapy); Part 2, Cohort B: Dose Expansion BMS-986497 (Triple Combination Therapy)
Drug: Venetoclax — Specified dose on specified days
  Arms: Part 2, Cohort B: Dose Expansion BMS-986497 (Triple Combination Therapy)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, drug levels, drug efficacy and determine the recommended dose of BMS-986497 as a monotherapy, in double combination with Azacitidine and in triple combination with Azacitidine and Venetoclax in participants with relapsed or refractory acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Adults with primary or secondary relapsed and/or refractory acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS).
* Detectable levels of cluster of differentiation 33 (CD33) expression.
* Failed alternative therapies with established benefit.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 and adequate organ function.

Exclusion Criteria:

* Acute Promyelocytic Leukemia.
* Clinically active central nervous system leukemia.
* Active malignant solid tumor.
* Pregnant or breastfeeding.
* Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2030-09-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to 21 days
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years
Determine the Recommended Phase 2 Dose (RP2D) of BMS-986497 as Monotherapy | Up to 2 years
RP2D of BMS-986497 as Combination Therapy | Up to 2 years
  The combination therapy included BMS-986497 and Azacitidine
RP2D of BMS-986497 as Triple Combination Therapy | Up to 2 years
  The triple combination therapy included BMS-986497, Azacitidine and Venetoclax.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Up to 2 years
Time to reach Cmax (Tmax) | Up to 2 years
Area under the curve from time 0 to last quantifiable concentration (AUC0-last) | Up to 2 years
Overall response rate (ORR) | Up to 4 years
Duration of response (DoR) | Up to 4 years
Best overall response (BOR) | Up to 4 years
Complete remission (CR) | Up to 4 years
Complete remission with incomplete hematologic recovery (Cri) | Up to 4 years
Complete remission with partial hematologic recovery (CRh) rate | Up to 4 years
Event-free survival (EFS) | Up to 4 years
Transition rate to allogeneic hematopoietic stem cell transplantation (HSCT) | Up to 4 years
Incidence of Anti-drug antibody (ADA) against BMS-986497 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (9):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Local Institution - 0007, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Local Institution - 0009, Fairfax, Virginia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (3):
  - Local Institution - 0017, Marseille, Bouches-du-Rhône
  - Local Institution - 0018, Paris
  - Local Institution - 0022, Toulouse
- Local Institution - 0020, Barcelona, Catalunya [Cataluña], Spain

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06419634.html